CLINICAL TRIAL: NCT04661423
Title: Use of RDS MultiSense® in Post-ICU Patients in the COVID-19 Era
Acronym: MONIREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Collaborators: Rhythm Diagnostic Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-004
Record Dates: First submitted 2020-12-07; First posted 2020-12-10 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Post ICU Rehabilitation
Keywords: Vital signs; Connected device; real-time monitoring; post-ICU; cardio-respiratory monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Remote Automated Monitoring System (Experimental): MultiSense® strip will be attached on patient's thorax. The monitoring will last between 5 and 7 days during the post-ICU hospitalization, at rest and during rehabilitation exercises.
  Interventions: Other: Remote Automated Monitoring System

INTERVENTIONS:
Other: Remote Automated Monitoring System — The patient will be monitored with conventional monitoring devices as well as the MultiSense patch.

SUMMARY:
In this clinical study, the investigators will compare vital parameters measurements obtained using continuous data from reference monitors and continuous wireless MultiSense® monitoring patch in 60 post-ICU (Intensive Care Unit) patients and over 7 days.

DETAILED DESCRIPTION:
The MultiSense® strip is a unique, band aid-sized, clinical signal quality, connected strip for real-time monitoring of cardio-respiratory parameters. The MultiSense® strip measures in real-time, remotely and continuously 11 clinical key-indicators by being attached to the patient thorax: ECG trace, heart rate, oxygen saturation (SpO2), respiratory rate and relative respiration depth, pulse transit time, plethysmographic trace, perfusion index, skin temperature, physical activity and body position. Designed to be worn continuously for at least seven days, the patient can keep the patch during his sleep or in the shower.

The aim of this study is to determine the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of accuracy, connectivity, generation of artifactual data and stability of data transmission. The study population includes 60 patients transferred to post-ICU units for a minimum of 5 days. Once in the post-ICU unit, the MultiSense® strip will be attached on patient's thorax. The monitoring will last between 5 to 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman over 18 years old.
* Patient previously cared in an ICU for severe COVID-19 pneumonia, COVID-related condition or similar neurological compromise necessitating post-ICU rehabilitation
* Negative respiratory SARS-CoV-2 (Severe Acute Respiratory Syndrome-Corona Virus-2) samples
* Patient admitted in a post-ICU rehabilitation unit with an expected length of stay > 5 days
* Patient able to receive and understand information related to the study and give written informed consent.

OR If the patient is not capable, presence of a next of kin able to receive and understand information related to the study and give written informed consent for the patient

* Patient authorizing the treatment of their personal data collected during the study (box checked in the consent form)
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patient with a skin disease that would preclude the use of an adhesive.
* Patient with an implantable device such as a pacemaker
* Pregnant or lactating patient.
* Patient in exclusion period (determined by a previous or a current study).
* Patient under guardianship or trusteeship.
* Patient under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-03-02 (Actual); Study Completion 2025-03-02 (Actual)

PRIMARY OUTCOMES:
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of accuracy. | from patch placement to hospital discharge, assessed up to 7 days
  Accuracy is defined as an average measurement variation less than 3.5 percent or 5 percent of the mean value, depending on the variable with respect to the reference standard.
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of connectivity. | from patch placement to hospital discharge, assessed up to 7 days
  Connectivity is defined as a time-wise ratio of missing versus total signal less than 20 percent.
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of generation of artifactual data. | from patch placement to hospital discharge, assessed up to 7 days
  The generation of artefact data is defined as a percentage of outlier data less than 10 percent.
Determination of the quality of measurements of clinical signs provided by MultiSense® strip in comparison to measurements made with conventional medical devices in the hospital setting, in terms of stability of data transmission. | from patch placement to hospital discharge, assessed up to 7 days
  Data transmission stability is defined as a data transmission rate equal to or greater than 80 percent.

SECONDARY OUTCOMES:
Usability of a data acquisition patch by health care providers (HCPs) in the setting of post-ICU, rehabilitation unit assessed via a questionnaire. | At hospital discharge, up to 7 days after the patch placement
  Descriptive determination of user-friendliness, comprehensibility and ease of placement, connection and removal of the data acquisition patch by healthcare providers.
User experience of post-ICU rehabilitation patients with the continuous use of the adhesive data acquisition patch during remote monitoring assessed via a patient's final questionnaire. | At hospital discharge, up to 7 days after the patch placement
  Descriptive determination of user experience and practicalities associated with wearing the data acquisition patch (e.g. portability, duration of skin adhesion, anticipated detachment, interference with activities and stigma perception).
Assess patients' tolerability to prolonged use of an adhesive patch during remote monitoring. | From patch placement to its removal (up to 7 days)
  Number of unexpected local and distant events attributable to the use of the adhesive data acquisition patch
Assess the correlation between body temperature and skin temperature | From patch placement to its removal (up to 7 days)
  Correlation between the body temperature measured with a standard device and the skin temperature measured with the remote data acquisition device.
Assess the ability of the patch to detect and signal the clinically confirmed excursions of heart rate (high and low) outside predefined thresholds | From patch placement to its removal (up to 7 days)
  Non-inferiority of the number of clinically confirmed alerts observed with the patch compared to those signalled by the conventional devices, and difference in the number of false positive excursions.
Assess the ability of the patch to detect and signal the clinically confirmed excursions of SpO2 (low) outside predefined thresholds | From patch placement to its removal (up to 7 days)
  Non-inferiority of the number of clinically confirmed alerts observed with the patch compared to those signalled by the conventional devices, and difference in the number of false positive excursions.
Assess the ability of the patch to detect and signal the clinically confirmed excursions of respiratory rate (high and low) outside predefined thresholds | From patch placement to its removal (up to 7 days)
  Non-inferiority of the number of clinically confirmed alerts observed with the patch compared to those signalled by the conventional devices, and difference in the number of false positive excursions.

CONTACTS AND LOCATIONS:
Overall Officials: Julien POTTECHER, MD, PhD, Principal Investigator — Anesthesia, Critical Care & Perioperative Medicine, Hautepierre, Strasbourg, France
Locations (2):
- France (2):
  - Anesthesia Department, Central Hospital, Nancy
  - Anesthesia, Critical Care & Perioperative Medicine, Hautepierre, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pamuk K, Turan N. The effect of light on sleep quality and physiological parameters in patients in the intensive care unit. Appl Nurs Res. 2022 Aug;66:151607. doi: 10.1016/j.apnr.2022.151607. Epub 2022 Jun 26. PMID 35840273